CLINICAL TRIAL: NCT01889394
Title: Primary Wound Closure Using a Limberg Flap Versus Secondary Wound Healing Following Pilonidal Sinus Excision: Short-term Results of a Randomized Controlled Multicenter Trial
Brief Title: Primary Wound Closure Using a Limberg Flap Versus Secondary Wound Healing Following Pilonidal Sinus Excision
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kantonsspital Liestal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UKBB 234/05
Record Dates: First submitted 2013-06-24; First posted 2013-06-28 (Estimated); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: Pilonidal Sinus
Keywords: pilonidal sinus; excision; primary wound closure; limberg flap
MeSH Terms: conditions — Pilonidal Sinus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- limberg flap (Active Comparator): primary wound closure using a limberg flap
  Interventions: Procedure: primary wound closure using a limberg flap
- secondary wound healing (Active Comparator): secondary wound healing
  Interventions: Procedure: secondary wound healing

INTERVENTIONS:
Procedure: secondary wound healing — secondary wound healing
  Arms: secondary wound healing
Procedure: primary wound closure using a limberg flap — primary wound closure using a limberg flap
  Arms: limberg flap

SUMMARY:
To compare primary wound closure using a limberg flap with secondary (p.s.) wound healing following excision of a pilonidal sinus.

DETAILED DESCRIPTION:
Patients who gave their informed consent who had excision of pilonidal sinus were randomly assigned to group A (primary wound closure with a Limberg flap) or to group B (open wound and p.s.wound healing).

ELIGIBILITY:
Inclusion Criteria:

* indication for excision of pilonidal sinus given

Exclusion Criteria:

* limberg flap not possible for surgical reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2006-01; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Inability to work | 1 year
  change for capacity for work at one year post-OP

SECONDARY OUTCOMES:
Pain perioperatively and after 3 weeks | 0 and 3 weeks
Complication rate after 3 weeks | 3 weeks
Patient satisfaction after 3 weeks & 1year | 3 weeks and 1 year
Recurrence rate after 1 year | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Christoph A Maurer, Prof Dr med, Principal Investigator — Department of General, Visceral, Vascular and Thoracic Surgery, Hospital of Liestal, Switzerland, affiliated with the University of Basel
Locations (3):
- Switzerland (3):
  - Kantonsspital Liest, Liestal, Basel-Landschaft
  - Gesundheitszentrum Fricktal, Rheinfelden, Canton of Aargau
  - Spitalzentrum Oberwallis, Visp, Valais